CLINICAL TRIAL: NCT04320316
Title: An Open Label Trial to Assess the Safety and Efficacy of KRN23, an Investigational Antibody to FGF23, in a Single Pediatric Patient With Epidermal Nevus Syndrome (ENS) and Associated Hypophosphatemic Rickets
Brief Title: A Trial to Assess the Safety and Efficacy of KRN23 in Epidermal Nevus Syndrome (ENS)
Acronym: ENS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Principal Investigator, Hussein D Abdullatif, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300004900
Record Dates: First submitted 2020-03-11; First posted 2020-03-25 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Epidermal Nevus Syndrome
Keywords: epidermal nevus syndrome; burosumab-twza
MeSH Terms: conditions — Nevus, Sebaceous of Jadassohn | interventions — burosumab; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crysvita (burosumab-twza) Treatment (Experimental): The starting dose will be 0.3 mg/kg to be given every 2 weeks. If required dose may be titrated with increments of 0.1 mg/kg/dose every 4 weeks up to a maximum of dose of 2.0mg/kg (not to exceed 90mg per dose) until phosphorus level is WNL.
  Patient will receive study drug via SC injection to the abdomen, upper arms, thighs, or buttocks; the injection site will be rotated with each injection. If the dose level exceeds 1.5 mL in volume, the dose should be administered at two injection sites.
  Duration of treatment is 52 weeks. Subjects that complete treatment through week 52 may have the option to continue KRN23 treatment. If this is warranted based on preliminary efficacy, the current protocol will be amended to allow for an extension.
  Interventions: Drug: Crysvita (burosumab-twza) Treatment

INTERVENTIONS:
Drug: Crysvita (burosumab-twza) Treatment — KRN23 is a fully human IgG1monoclonal antibody that binds to and inhibits the activity of FGF23, leading to an increase in serum phosphorus levels. It is a potential therapeutic candidate for the treatment of XLH, Tumor-Induced Osteomalacia (TIO), and the rickets/osteomalacia resulting from Epidermal Nevus Syndrome (ENS). All of these conditions are diseases of bone hypomineralization, caused by urinary phosphate wasting due to elevated levels of FGF23.
  Other Names: no other names available

SUMMARY:
KRN23 is a fully human immunoglobulin monoclonal antibody (mAb) that binds to and inhibits the activity of fibroblast growth factor 23 (FGF23), leading to an increase in serum phosphorus levels. There are multiple disorders that result in unusually high circulating levels of FGF23, which in turn result in renal phosphate wasting and reduced levels of 1,25-dihydroxy vitamin D (1,25[OH]2D). Across these disorders the clinical symptoms are similar and often include osteomalacia (and, in children, rickets), muscle weakness, fatigue, bone pain, and fractures. KRN23 has been studied in one of these disorders, X-linked hypophosphatemia (XLH). In single- and repeat-dose clinical studies in subjects with XLH, subcutaneous (SC) administration of KRN23 consistently increased and sustained serum phosphorus levels and tubular reabsorption of phosphate (TRP) without a major impact on urine calcium levels or vitamin D metabolism. Positive results were also observed in a nonclinical pharmacology model of XLH. It is hypothesized that KRN23 may provide clinical benefit in this patient due to the common underlying feature in this patient and in patients with XLH - abnormally elevated FGF23 in the context of low age -adjusted serum phosphorous levels. The primary objective is to study the effect of KRN23 treatment on normalizing age-adjusted fasting serum phosphorous levels in a single pediatric patient with Epidermal Nevus Syndrome associated hypophosphatemic rickets.

DETAILED DESCRIPTION:
KRN23 is a fully human immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that binds to and inhibits the activity of fibroblast growth factor 23 (FGF23), leading to an increase in serum phosphorus levels. There are multiple disorders (each with a unique underlying cause) that result in unusually high circulating levels of FGF23, which in turn result in renal phosphate wasting and reduced (or aberrantly normal in relationship to elevated FGF23) levels of 1,25-dihydroxy vitamin D (1,25[OH]2D). Across these disorders the clinical symptoms are similar and often include osteomalacia (and, in children, rickets), muscle weakness, fatigue, bone pain, and fractures. KRN23 has been studied in one of these disorders, X-linked hypophosphatemia (XLH). In single- and repeat-dose clinical studies in subjects with XLH, subcutaneous (SC) administration of KRN23 consistently increased and sustained serum phosphorus levels and tubular reabsorption of phosphate (TRP) without a major impact on urine calcium levels or vitamin D metabolism. Positive results were also observed in a nonclinical pharmacology model of XLH. It is hypothesized that KRN23 may provide clinical benefit in this patient due to the common underlying feature in this patient and in patients with XLH - abnormally elevated FGF23 in the context of low age -adjusted serum phosphorous levels.

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed ENS by physician diagnosis
* Patient has confirmed FGF23 elevations in the context of low serum phosphorous < 4.1 mg/dL
* Patient able to tolerate KRN23 treatment
* Have a corrected serum calcium level < 10.8mg/dL
* Have an eGFR >60 ml/min
* Must be willing in the opinion of the investigator, to comply with study procedures and schedule
* Provide written informed consent by a parent after

Exclusion Criteria:

* Patient should not use CRYSVITA with Oral phosphate or active Vitamin D analogs.
* Patient and investigator should not initiate CRYSVITA if Phosphorus level is within or above normal.
* CRYSVITA is contraindicated in patients with severe renal impairment or end stage renal disease because these conditions are associated with abnormal mineral metabolism.
* The use or enrollment in studies using other investigational therapies including other monoclonal antibodies
* Subject and their Parent not willing or not able to give written informed consent
* In the Investigators opinion, the subject may not be able to meet all the requirements for study participation
* Subject has a history of hypersensitivity to KRN23 excipients that in the opinion of the investigator, places the subject at an increased risk of adverse effects
* Subject has a condition that in the opinion of the investigator could present a concern for subject safety or data interpretation.

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Abdul-Latif, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Derived] Huynh C, Gillis A, Fazendin J, Abdullatif H. A case report to assess the safety and efficacy of Burosumab, an investigational antibody to FGF23, in a single pediatric patient with Epidermal Nevus Syndrome and associated hypophosphatemic rickets. Bone Rep. 2022 Jul 20;17:101605. doi: 10.1016/j.bonr.2022.101605. eCollection 2022 Dec. PMID 35899095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited 1 patient with Epidermal nevus and hypophosphatemia
Groups:
- Crysvita (Burosumab-twza) Treatment: The starting dose will be 0.3 mg/kg to be given every 2 weeks. If required dose may be titrated with increments of 0.1 mg/kg/dose every 4 weeks up to a maximum of dose of 2.0mg/kg (not to exceed 90mg per dose) until phosphorus level is WNL.
  Patient will receive study drug via SC injection to the abdomen, upper arms, thighs, or buttocks; the injection site will be rotated with each injection. If the dose level exceeds 1.5 mL in volume, the dose should be administered at two injection sites.
  Duration of treatment is 52 weeks. Subjects that complete treatment through week 52 may have the option to continue KRN23 treatment. If this is warranted based on preliminary efficacy, the current protocol will be amended to allow for an extension.
  Crysvita (burosumab-twza) Treatment: KRN23 is a fully human IgG1monoclonal antibody that binds to and inhibits the activity of FGF23, leading to an increase in serum phosphorus levels. It is a potential therapeutic candidate for the treatment of XLH, Tumor-Induced Osteomalacia (TIO), and the rickets/osteomalacia resulting from Epidermal Nevus Syndrome (ENS). All of these conditions are diseases of bone hypomineralization, caused by urinary phosphate wasting due to elevated levels of FGF23.
Period: Overall Study
Arm/Group | Crysvita (Burosumab-twza) Treatment
Started (Patient started on Burosumab and the dose was adjusted upwards every 4 weeks because of still having relatively low Phsophorus level.) | 1 (1)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: people with Epidermal nevus and also hypophopshatemia.
Groups:
- Crysvita (Burosumab-twza) Treatment: The starting dose will be 0.3 mg/kg to be given every 2 weeks. If required dose may be titrated with increments of 0.1 mg/kg/dose every 4 weeks up to a maximum of dose of 2.0mg/kg (not to exceed 90mg per dose) until phosphorus level is WNL.
  Patient will receive study drug via SC injection to the abdomen, upper arms, thighs, or buttocks; the injection site will be rotated with each injection. If the dose level exceeds 1.5 mL in volume, the dose should be administered at two injection sites.
  Duration of treatment is 52 weeks. Subjects that complete treatment through week 52 may have the option to continue KRN23 treatment. If this is warranted based on preliminary efficacy, the current protocol will be amended to allow for an extension.
  Crysvita (burosumab-twza) Treatment: KRN23 is a fully human IgG1monoclonal antibody that binds to and inhibits the activity of FGF23, leading to an increase in serum phosphorus levels. It is a potential therapeutic candidate for the treatment of XLH, Tumor-Induced Osteomalacia (TIO), and the rickets/osteomalacia resulting from Epidermal Nevus Syndrome (ENS). All of these conditions are diseases of bone hypomineralization, caused by urinary phosphate wasting due to elevated levels of FGF23.
  The primary measure of the study is to see a rise of the phosphorus level to the normal range or as close as possible to the normal range.
Arm/Group | Crysvita (Burosumab-twza) Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Participant Will Achieve Normal Age-adjusted Phosphorous Levels as Tested by Fasting Serum Lab Values
Description: Checking PO4 levels every two weeks and adjusting doses every 4 weeks in blood
Time Frame: every 2 week, from baseline to 52 weeks.
Population: Same as above with only 1 patient
Measure: Number; unit: mg/dl
Arm/Group | Crysvita (Burosumab-twza) Treatment
Number analyzed (Participants) | 1
mg/dl
  baseline | 0.8
  2 week | 1.2
  4 week | 1.3
  6 week | 1.1
  8 week | 1.4
  10 week | 1.7
  12 week | 1.9
  14 week | 1.3
  16 week | 2
  18 week | 2.3
  20 week | 1.8
  22 week | 2.1
  24 week | 2.1
  26 week | 2.3
  28 week | 2.6
  30 week | 2
  32 week | 1.9
  34 week | 1.8
  36 week | 2.1
  38 week | 2.5
  40 week | 2.9
  42 weeks | 2.7
  44 weeks | 1.8
  46 week | 2.4
  48 weeks | 2.6
  50 | 2.5
  52 | 3.3

2. Secondary Outcome: Participant Will Achieve Improving Vitamin D Levels as Measured by Serum Blood Tests.
Description: check Vitamin D 1,25 in blood every 3 months
Time Frame: 1 year
Population: one patient with Epidermal nevus and hypophosphatemia
Measure: Number; unit: pg/ml
Groups:
- Vitamin D Level on Treatment: obtain levels of Vitamin D 1,25 in blood
Arm/Group | Vitamin D Level on Treatment
Number analyzed (Participants) | 1
pg/ml
  Baseline Vit D 1,25 | 15
  2 months Vit D 1,25 | 68
  6 months Vit D 1,25 | 105
  9 months Vita D 1,25 | 95
  1 year Vit D 1,25 | 115

3. Secondary Outcome: Participant Will Achieve Improving iPTH Levels as Measured by Serum Blood Tests.
Description: measure PTH levels approximately every 3 months
Time Frame: every 3 months, From Baseline to 52 weeks
Population: same as above
Measure: Number; unit: pg/ml
Groups:
- PTH Levels: obtain blood levels of parathyroid hormone (PTH)
Arm/Group | PTH Levels
Number analyzed (Participants) | 1
pg/ml
  baseline PTH | 334.5
  3 months | 334.1
  6 months | 317
  9 months | 245.9
  1 year | 330.4

4. Secondary Outcome: Participant Will Achieve Improving Calcium Levels as Measured by Serum Blood Tests.
Description: measure Calcium level every 3 months
Time Frame: every 3 months, From Baseline to 52 weeks
Population: same as above
Measure: Number; unit: mg/dl
Groups:
- Calcium Levels: taking blood calcium level
Arm/Group | Calcium Levels
Number analyzed (Participants) | 1
mg/dl
  baseline Calcium | 10.5
  3 months | 10.5
  6 months | 11.2
  9 months | 12
  1 year | 13.4

5. Secondary Outcome: Participant Will Achieve Improvement of Underlying Skeletal Disease/Rickets as Assessed by Standard Radiographs.
Description: DEXA (dual energy X-ray Absorbometry) scans and whole body x-rays will be taken at baseline. A lower Z score is indicative of poor results. Z score compares the standard deviations of the reading with matched aged persons. The normal range is +2 to - 2 Standard deviations and those are what we call Z scores. A Z score of 0 is the population mean.
Time Frame: baseline scans prior to drug administration
Population: same as above
Measure: Number; unit: Z score
Groups:
- DEXA Scan: DEXA scan was obtained at baseline. A DEXA scan is a bone densitometry measure.
Arm/Group | DEXA Scan
Number analyzed (Participants) | 1
Z score | -3.9

6. Secondary Outcome: Participant Will Achieve Improving Levels of Alkaline Phosphatase (ALP)
Description: obtain Alkaline phosphatase in blood every 3 months
Time Frame: every 3 months, From baseline to 52 weeks
Population: same as above
Measure: Number; unit: U/L
Groups:
- Alkaline Phosphatase: The Alkaline phosphatase is measured in blood every 3 months. it is a measure of bone activity.
Arm/Group | Alkaline Phosphatase
Number analyzed (Participants) | 1
U/L
  baseline | 672.4
  3 months | 468.3
  6 months | 313
  9 months | 287
  1 year | 185.2

ADVERSE EVENTS:
Time Frame: 1 year
Description: No serious adverse events occurred
Groups:
- Adverse Events: No adverse events occurred. Adverse events were not monitored/collected by dose level.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The patient is wheel chair bound and so we could not obtain data on mobility before or after the trial. We were not able to check a DEXA scan at the end of the study either.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04320316/Prot_SAP_001.pdf